CLINICAL TRIAL: NCT03394664
Title: Macronutrients and Body Fat Accumulation: A Mechanistic Feeding Study
Brief Title: FB4 (Framingham, Boston, Bloomington, Birmingham, and Baylor)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The FB4 trial has been terminated due to COVID-19.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Indiana University (Other); University of Alabama at Birmingham (Other); Framingham State University (Other); Baylor University (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Co-Director, New Balance Foundation Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00026977
Record Dates: First submitted 2017-12-29; First posted 2018-01-09 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Body composition; Feeding study; Ketogenic diet; Weight loss; Energy Expenditure
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors conducting analyses of biospecimens, laboratory personnel, DXA technologists, and research nurses were blinded to random group assignment. They were not involved in the randomization process or any aspects of the intervention. The statistical team worked with masked labels for the diet arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Very-Low Carbohydrate Diet (Experimental): Feeding study. Dietary composition (approximately): 75% fat
  Interventions: Behavioral: Feeding Study
- High-Carbohydrate Low-Sugar Diet (Experimental): Feeding study. Dietary composition (approximately): 25% fat 0% added sugars.
  Interventions: Behavioral: Feeding Study
- High-Carbohydrate High-Sugar Diet (Experimental): Feeding study. Dietary composition (approximately): 25% fat, 20% added sugars.
  Interventions: Behavioral: Feeding Study

INTERVENTIONS:
Behavioral: Feeding Study — Food provision throughout the study: 1) Run-In Phase (VLC diet, weight loss); 2) Residential Phase (3 different test diets, weight-loss maintenance).
  Other Names: weight loss, weight-loss maintenance

SUMMARY:
This study will evaluate the effects of dietary carbohydrate and sugar consumption, independent of energy content, on body fatness and metabolism in a rigorous feeding study.

DETAILED DESCRIPTION:
Many people with obesity can lose weight for a few months, but most have difficulty maintaining weight loss over the long term. Extensive research has shown that weight loss elicits biological adaptations - including a decline in energy expenditure and an increase in hunger - that promote weight regain. However, this observation leaves unanswered why average body weight has recently increased among populations that are mostly genetically stable. According to the Carbohydrate-Insulin Model, increased consumption of processed carbohydrates during the low-fat diet era of the last 40 years has raised the average body weight being defended by biological mechanisms on a population basis. Specifically, the investigators hypothesize that diets high in total carbohydrate (with or without added sugar) acting through increased insulin secretion, alter substrate partitioning toward storage in body fat, leading to increased hunger, slowing metabolism, and accumulation of body fat.

To test this hypothesis, the investigators plan a randomized-controlled feeding study involving 125 adults with obesity. During the run-in phase, participants will be given a hypocaloric very-low-carbohydrate (VLC) diet, with adjustment of energy intake to produce 15 ± 3% weight loss over 3 to 4 months on an outpatient basis. After weight stabilization, participants will be admitted to a residential center for 13 weeks. During the first 3 weeks, energy intake and expenditure will be closely monitored during weight-loss maintenance. Then, energy intake will be individually "locked" at levels equal to energy expenditure and participants will be administered one of three randomly-assigned test diets for 10 weeks. The test diets include VLC, High Carbohydrate-Low Sugar (HC-LS), and High Carbohydrate-High Sugar (HC-HS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years
* BMI ≥ 27 kg/m2
* Weight ≤ 350 lb
* Medical clearance from a primary care provider
* Willingness to follow a VLC weight-loss diet
* Willingness to reside in a research unit for 3 months and eat/drink only provided study foods and beverages
* No major food allergies or aversions
* Willingness to obtain seasonal flu shot or provide documentation of flu shot for current flu season (winter/spring cohort only)
* Willingness to discuss work options (e.g., remote work) with employer, and make appropriate arrangements prior to the Residential phase.

Exclusion Criteria:

* Change in body weight ≥ 10% during prior 6 months
* Specialized diets (e.g., for medical or religious reasons)
* Chronic use of any medication or dietary supplement that could affect study outcomes (e.g., insulin, metformin, thyroxine)
* Current smoking (1 cigarette in the last week)
* Greater than moderate alcohol consumption (> 14 drinks/wk) or history of binge drinking (≥5 drinks in 1 day within past 6 months)
* Physician diagnosis of a major medical illness or eating disorder
* History of kidney stones
* Laboratory tests: ALT>2x upper limit; abnormal HgA1c; abnormal TSH; abnormal creatinine; abnormal uric acid (using the male upper limit for both sexes)
* Failed criminal offender background check or sex offender background check
* Use of recreational drugs
* Current diagnosis or history of kidney stones, gout, or gall stones; or removal of gall bladder
* Exercise restrictions or at high risk for complications during exercise

Female-specific exclusion criteria:

* Menopausal
* Any change in birth control medication during the 3 months prior to enrollment
* Pregnancy or lactation during the 12 months prior to enrollment, or intent to become pregnant during study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Body fat mass | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Body composition assessed using a multi-component model

SECONDARY OUTCOMES:
Lean body mass | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed using a multi-component model (difference between total body mass and fat mass)
Body weight | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Anthropometrics, assessed by calibrated scale, in kilograms (kg)
Total energy expenditure (TEE) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed using doubly labeled water methodology
Resting energy expenditure (REE) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by indirect calorimetry using respiratory gas exchange methodology with a ventilated hood system
Physical activity level, (moderate to vigorous) | Measurements made daily during 2 weeks at PWL, 2 weeks at END, and alternating non-assessment weeks of the residential phase and integrated into a unified outcome
  Total minutes of moderate- to vigorous-intensity physical activity, assessed by accelerometry
Insulin sensitivity | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by frequently-sampled oral glucose tolerance test [OGTT], calculated using plasma insulin and glucose values
Insulin secretion | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by frequently-sampled oral glucose tolerance test [OGTT], using plasma insulin at 30 minutes following the dose of dextrose
Glycemic control | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Hemoglobin A1c [HbA1c]
Total cholesterol | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Chronic disease risk factor
HDL-cholesterol | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Chronic disease risk factor
LDL-cholesterol | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Chronic disease risk factor
Non-HDL cholesterol | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Chronic disease risk factor
Triglycerides | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Chronic disease risk factor
Plasminogen Activator Inhibitor-1 [PAI-1] | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Indicator of coagulopathy
High-sensitivity C-reactive protein [hsCRP] | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Indicator of chronic inflammation
Uric acid | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Indicator of risk for kidney stones, measured in blood
Systolic blood pressure | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by auscultation, mmHg
Diastolic blood pressure | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by auscultation, mmHg
Thyroxine (T4) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Thyroid function
Free T4 | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Thyroid function
Thyroid stimulating hormone [TSH] | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Thyroid function
Insulin-like growth factor-1 [IGF-1] | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Growth hormone action
Urine cortisol | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Stress hormone, assessed using 24-hour urine collection
Urine catecholamines | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Stress hormone, assessed using 24-hour urine collection
Leptin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Adipokine
Total Adiponectin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Adipokine
High-molecular weight adiponectin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Adipokine
Sleep | Measurements made daily during 2 weeks at PWL, 2 weeks at END, and alternating non-assessment weeks of the residential phase and integrated into a unified outcome
  Total sleep time, sleep onset latency, wake after sleep onset, and sleep efficiency, assessed by accelerometry
Blood glucose | Measurements made daily during residential phase (0 to 10 weeks) and integrated into a unified outcome
  Assessed by continuous glucose monitoring (CGM)
Ghrelin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Hormonal Control of Appetite
Body Circumference | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed using a 3D body scan
Post-prandial energy expenditure and respiratory quotient | Single assessment in weeks 6 to 8 of residential study
  Optional testing, assessed by indirect calorimetry using respiratory gas exchange
Activation of insulin signaling pathways | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Assessed by immunohistochemistry of phosphorylated insulin receptor and signaling proteins

OTHER OUTCOMES:
1,5-anhydroglucitol (1,5-AG) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Lipoprotein particle subfraction distribution | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Fibrinogen | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Interleukin-6 (IL-6) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Reverse triiodothyronine (rT3) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Insulin-like growth factor-binding protein 3 (IGF-BP3) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Luteinizing hormone (LH) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Follicle stimulating hormone (FSH) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Estradiol (E2) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Testosterone (TST, total) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Testosterone (TST, free) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Metabolomics profile | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Biomarker of cholesterol synthesis | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Biomarker of cholesterol absorption | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
MicroRNA | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Gut microbiome | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived specimen
Demographics (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Body composition (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Measure of glucose homeostasis (insulin-30) (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Measure of glucose homeostasis (insulin sensitivity) (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Measure of glucose homeostasis (glycemic control) (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Obesity related genetic risk (mediator/modifier) | Pre-weight loss baseline
  Baseline covariate
Body composition (mediator/modifier) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Time varying covariate
Measure of glucose homeostasis (insulin-30) (mediator/modifier) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Time varying covariate
Measure of glucose homeostasis (insulin sensitivity) (mediator/modifier) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Time varying covariate
Measure of glucose homeostasis (glycemic control) (mediator/modifier) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Time varying covariate
Physical activity level (moderate to vigorous) (mediator/modifier) | Measurements made daily during 2 weeks at PWL, 2 weeks at END, and alternating non-assessment weeks of the residential phase and integrated into a unified outcome
  Time varying covariate for total minutes of moderate to vigorous intensity physical activity, assessed by accelerometry.
Sex Hormone-Binding Globulin (SHBG) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analysis of archived specimen
Urinary nitrogen | End of residential (END, 10 weeks)
  Archived for future analysis
Glucagon-like peptide-1 (GLP-1) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived samples
Glucose-dependent insulinotropic polypeptide (GIP) | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived samples
Glucagon | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived samples
Oxytocin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived samples
Oxyntomodulin | Change from post-weight loss (PWL, 0 weeks) to end of residential study (END, 10 weeks)
  Possible future analyses of archived samples

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; David B Allison, PhD, Principal Investigator — Indiana University, Bloomington; Cara B Ebbeling, PhD, Study Director — Boston Children's Hospital
Locations (1):
- Warren Conference Center and Inn, Ashland, Massachusetts, United States

REFERENCES:
- [Background] Ludwig DS, Friedman MI. Increasing adiposity: consequence or cause of overeating? JAMA. 2014 Jun 4;311(21):2167-8. doi: 10.1001/jama.2014.4133. No abstract available. PMID 24839118
- [Background] Ebbeling CB, Swain JF, Feldman HA, Wong WW, Hachey DL, Garcia-Lago E, Ludwig DS. Effects of dietary composition on energy expenditure during weight-loss maintenance. JAMA. 2012 Jun 27;307(24):2627-34. doi: 10.1001/jama.2012.6607. PMID 22735432
- [Derived] Wong MC, Bennett JP, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Wong JMW, Ebbeling CB, Ludwig DS, Irving BA, Scott MC, Stampley J, Davis B, Johannsen N, Matthews R, Vincellette C, Garber AK, Maskarinec G, Weiss E, Rood J, Varanoske AN, Pasiakos SM, Heymsfield SB, Shepherd JA. Monitoring body composition change for intervention studies with advancing 3D optical imaging technology in comparison to dual-energy X-ray absorptiometry. Am J Clin Nutr. 2023 Apr;117(4):802-813. doi: 10.1016/j.ajcnut.2023.02.006. Epub 2023 Feb 14. PMID 36796647
- [Derived] Jansen LT, Yang N, Wong JMW, Mehta T, Allison DB, Ludwig DS, Ebbeling CB. Prolonged Glycemic Adaptation Following Transition From a Low- to High-Carbohydrate Diet: A Randomized Controlled Feeding Trial. Diabetes Care. 2022 Mar 1;45(3):576-584. doi: 10.2337/dc21-1970. PMID 35108378
- [Derived] Wong JMW, Yu S, Ma C, Mehta T, Dickinson SL, Allison DB, Heymsfield SB, Ebbeling CB, Ludwig DS. Stimulated Insulin Secretion Predicts Changes in Body Composition Following Weight Loss in Adults with High BMI. J Nutr. 2022 Mar 3;152(3):655-662. doi: 10.1093/jn/nxab315. PMID 34587231